CLINICAL TRIAL: NCT07323030
Title: COMPARISON OF TWO DIFFERENT THERAPEUTIC ULTRASOUND TECHNIQUES IN COMBINATION WITH STANDARD PHYSICAL THERAPY VERSUS STANDARD PHYSICAL THERAPY ALONE IN PATIENTS WITH KNEE OSTEOARTHRITIS
Brief Title: THERAPEUTIC ULTRASOUND IN PATIENTS WITH KNEE OSTEOARTHRITIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Dilek ün oguzhanasilturk, Physical Medicine and Rehabilitation Specialits, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: okm-230
Record Dates: First submitted 2025-12-21; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Knee Osteoarthritis
Keywords: Therapeutic ultrasound; Physical Therapy; Ultrasound application techniques; Knee pain; Functional outcome
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: This is prosrective ,parallel group interventional study evaluating the effectiveness of therapeutic ultrasound in patients with gonartrosis
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- continius ultrasound group (Experimental): hot pack,tens,exercise terapy ,continius ultasound
  Interventions: Device: hot pack; Device: transcutaneus electrical nerve stimulatıon; Behavioral: exersice terapy; Device: continius ultrasound
- pulse ultrasound group (Experimental): hot pack,tens,exercise terapy,pulsed ultrasound
  Interventions: Device: hot pack; Device: transcutaneus electrical nerve stimulatıon; Behavioral: exersice terapy; Device: pulsed ultrasound
- control group (Experimental): hot pack,tens,exercise terapy
  Interventions: Device: hot pack; Device: transcutaneus electrical nerve stimulatıon; Behavioral: exersice terapy

INTERVENTIONS:
Device: hot pack — superficial heat therapy applied to the knee joınt using hot packs before other pyhsical terapy modalites .Hot packs are applied for approximately 15-20 minutes per session
Device: transcutaneus electrical nerve stimulatıon — TENS is a non-invasive electrical stimulation technique applied through surface electrodes to modulate sensory nerve activity without producing muscle contraction.
Behavioral: exersice terapy — Exercise therapy is a structured, planned, and repetitive physical intervention designed to improve or maintain physical function, mobility, strength, balance, and overall health through targeted therapeutic exercises.
Device: continius ultrasound — Continuous ultrasound is a therapeutic modality in which high-frequency sound waves are delivered continuously to biological tissues to produce predominantly thermal effects, leading to increased tissue temperature, enhanced blood flow, improved tissue extensibility, and pain modulation.
  Arms: continius ultrasound group
Device: pulsed ultrasound — Pulsed ultrasound is a therapeutic ultrasound modality in which acoustic energy is delivered intermittently rather than continuously, resulting in predominantly non-thermal mechanical effects such as cavitation and acoustic microstreaming that promote tissue healing and reduce inflammation.
  Arms: pulse ultrasound group

SUMMARY:
Knee osteoarthritis is a common condition that causes pain, stiffness, and reduced physical function. Therapeutic ultrasound is frequently used in physical medicine and rehabilitation to reduce pain and improve joint function in patients with knee osteoarthritis; however, different ultrasound application techniques are used in clinical practice.

The aim of this study was to compare the effectiveness of two different therapeutic ultrasound techniques in patients with knee osteoarthritis. Participants with knee osteoarthritis received therapeutic ultrasound treatment using one of two application techniques according to a predefined treatment protocol. Clinical outcomes related to pain and functional status were evaluated before and after treatment.

This completed study provides information on whether different ultrasound application techniques lead to differences in clinical outcomes in patients with knee osteoarthritis and may help guide clinical decision-making in rehabilitation practice.

DETAILED DESCRIPTION:
This study was designed as a prospective, parallel-group interventional study to evaluate the clinical effectiveness of different therapeutic ultrasound application techniques in patients diagnosed with knee osteoarthritis.

Eligible participants with knee osteoarthritis were allocated into treatment groups according to the predefined study protocol. Therapeutic ultrasound was applied using two different techniques under standardized treatment parameters. All participants received treatment sessions over a defined treatment period.

Clinical outcome measures related to pain intensity and functional status were assessed at baseline and after completion of the treatment protocol. Outcome assessments were performed by an evaluator blinded to group allocation.

The primary objective of the study was to compare the effects of different therapeutic ultrasound techniques on pain reduction and functional improvement in patients with knee osteoarthritis. Secondary objectives included evaluating changes in physical function following treatment.

ELIGIBILITY:
Inclusion Criteria:

Age between 40 and 75 years,Clınıcal and radıografıc dıagnosısı of knee osteoartrıtsı accordıng to Amerıcan College of Rheumatology crıteria,Kellegren Lawrencw grade 2-3 osteoartritis,prencense of knee pain for at least 3 months,ability to ambulate independently, ability to understand and comply with study procedures

Exclusion Criteria:

* History of knee surgery or ıntraartıkuler ınjection within the 6 last month,severe knee osteoaertırtıcs (kellegren lawrence grade 4),Neurological disorders affecting lower exremity functıon ,pulmoner or systemic disease limitin participitian,pregnancy,current partpiciant ın another clinical trial

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
pain intensity assessed by visuel analog scale (VAS) | baseline,immediately after treatment, and 2 months post-tratment
  Pain intensity was assessed using a 10-cm visual analog scale (VAS), where 0 indicates no pain and 10 indicates the worst imaginable pain. Participants marked their perceived knee pain level at each assessment point.
knee joint stiffness assessed by WOMAC stiffness subscale | baseline,immediately after treatment and at 2 months post treatment
  Knee joint stiffness was evaluated using the stiffness subscale of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). Higher scores indicate greater stiffness and symptom severity.
lesquesne algofunctional ındex score | baseline,immediately after treatment,and at 2 months post-treatment
  Functional impairment related to knee osteoarthritis was assessed using the Lequesne algofunctional index, which evaluates pain, walking distance, and activities of daily living. Higher scores reflect greater functional disability.

SECONDARY OUTCOMES:
Quadriceps muscle strength assesed by isokinetic dynamometry | baseline,immediately after treatment and 2 monthspost treatment
  Quadriceps muscle strength was measured using isokinetic dynamometry under standardized testing conditions. Peak torque values were recorded to assess muscle strength performance.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Ün oguzhanasiltürk, Principal Investigator — Kanuni Sultan and Süleyman Training Resarch Hospital
Locations (1):
- Prof .Dr .Cemil Taşcioğlu City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
İndividual participipant data will not be shared,as data sharing was not included in the study protocol and ethics committee approval ,and paricipant confidentiality must be maintained.